CLINICAL TRIAL: NCT00914810
Title: Effect of Supplemental Vitamin D on Skeletal Muscle Function in COPD Patients.
Brief Title: Effect of Supplemental Vitamin D on Skeletal Muscle Function in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ken M. Kunisaki, Assistant Professor of Medicine and Staff Physician, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4129-A
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; Vitamin D; Cholecalciferol; Skeletal muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Cholecalciferol (2000 I.U. daily)
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- Placebo (Placebo Comparator): Placebo capsule (sugar pill daily)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — 2000 I.U. daily for 6 weeks
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo (sugar pill) daily for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether or not vitamin D supplementation can improve physical performance in persons with severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Forced expiratory volume in one second (FEV1) < or = 50% of predicted
* Smoking history of at least 10 pack-years
* Able to ambulate independently or with the use of an ambulatory assist device (such as a cane or walker)

Exclusion Criteria:

* Currently taking > 500 I.U. per day of vitamin D supplements
* Primary diagnosis of asthma
* Uncompensated heart failure
* Heart attack in the previous 6 months
* Kidney disease (glomerular filtration rate < 45 mL/min/1.73m2)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken M. Kunisaki, M.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the Minneapolis Veterans Affairs Health Care System were recruited as a convenience sample between January 2009 and October 2011 from outpatient pulmonary clinics and an institutional review board-approved database of patients with COPD.
Groups:
- Placebo: Placebo : Placebo (sugar pill) daily for 6 weeks
- Vitamin D: Vitamin D (cholecalciferol) : 2000 I.U. daily for 6 weeks
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 20 | 19
Completed | 18 | 18
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Relocated out of state | 1 | 0
Not completed — Hospitalized and unable to follow up. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 20 | 19 | 39
Age Continuous [Mean (Standard Deviation); unit: years]
  Age | 68 (8) | 67.6 (7) | 68 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Physical Performance Battery (SPPB) Score
Description: SPPB measures lower extremity strength using 3 simple office-based tests to assess standing balance, gait speed, and chair stands. The composite SPPB score ranges from 0 (worst performance) to 12 (best performance). The minimal clinically important difference is not fully agreed upon, although a difference of 1.0 point has been used in many studies.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 18 | 18
units on a scale | 0.6 (1.7) | 0.9 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority or Other; p = 0.55, t-test, 2 sided; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.8 to 1.5]

2. Secondary Outcome: Change in Blood Level of Vitamin D (25-hydroxyvitamin D)
Time Frame: Baseline and 6 weeks
Population: 25-hydroxyvitamin D levels missing for 2 participants in the vitamin D arm of the trial.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 18 | 16
ng/mL | -1.8 (3.1) | 8.7 (5.5)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 10.5, 95% CI 2-sided [7.4 to 13.6]

ADVERSE EVENTS:
Arm/Group | Placebo | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No